CLINICAL TRIAL: NCT01332747
Title: Clinical Study on Hyperlipidemia and Comparative Evaluation of Efficacy of a Compound Unani Formulation (Safoof e Muhazzil) and Compressed Tablet of Safoof e Muhazzil in Its Management
Brief Title: Clinical Study to Evaluate Antihyperlipidemic Effect of a Classical Unani Antiobesity Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jamia Hamdard University (Other)
Responsible Party: Principal Investigator, Umar Jahangir, Lecturer, Jamia Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD/SM/2008-11
Record Dates: First submitted 2011-04-05; First posted 2011-04-11 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Hyperlipidemia
Keywords: TC; TG; HDL; LDL; VLDL
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Safoof e Muhazzil in its conventional powder form (Experimental): safoof e muhazzil in its conventional powder form 5 gms twice daily given orally
  Interventions: Drug: safoof e muhazzil
- compressed tablet of safoof e muhazzil (Experimental): compressed tablet of safoof e muhazzil is given in equivalent dose orally
  Interventions: Drug: compressed tablet of safoof e muhazzil
- atorvastatin (Active Comparator): atorvastatin 10mg daily as a standard control
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: safoof e muhazzil — drug is composed of 5 herbal(Carum Carvi,Trachyspermum copticum,Foeniculum Vulgare,Origanum Vulgare,Ruta Graveolens) 1 animal origin (Lac)and 1 mineral origin (Borax) ingredients.
  to be given in a dosage of 5 gms twice daily
  Arms: Safoof e Muhazzil in its conventional powder form
Drug: compressed tablet of safoof e muhazzil — drug is composed of 5 herbal(Carum Carvi,Trachyspermum copticum,Foeniculum Vulgare,Origanum Vulgare,Ruta Graveolens) 1 animal origin (Lac)and 1 mineral origin (Borax) ingredients.
  compressed into tablets of 1 gm each+ binders qs. dose is 5 tablets twice daily
  Arms: compressed tablet of safoof e muhazzil
Drug: Atorvastatin — atorvastatin 10 mgs once daily
  Arms: atorvastatin

SUMMARY:
The purpose of this clinical trial is to study the comparative effect of a classical unani antiobesity drug safoof-e-muhazzil on hyperlipidemia in its classical powder form and in compressed tablet form against a standard control.

DETAILED DESCRIPTION:
* The largest proportion of cardiovascular diseases is represented by Coronary artery disease(CAD), cerebral and peripheral vascular diseases. During the past decades efficacious strategies have been developed for prevention of these diseases. These strategies involve general lifestyle changes, which include, healthy diet, optimal weight, physical activity, moderate or no alcohol consumption, and smoking cessation, treatment of high blood pressure, control of diabetes mellitus and in particular, treatment of hyperlipidemia.
* Major clinical trials carried out, have shown a clear benefit of low density lipoprotein-cholesterol(LDL-C) reduction in terms of both CAD events and total mortality. A similar reduction in the relative risk of coronary events has been documented in patients with and without clinically evident CAD and in patients with mild or severe hyperlipidemia.
* Hyperlipidemia can be primary which is gene related causing defects in the synthesis of lipoprotein degradation. The other type of hyperlipidemia is secondary which is subsequent to related metabolic abnormalities.
* Although several Unani physicians have mentioned considerable details about fats in blood but it is observed that Hyperlipidemia has not been mentioned per se in the classical Unani literature.
* A condition that resembles hyperlipidemia in various aspects like etiology, clinical features and complications has been described as obesity in the classical Unani literature and mentions related methods for managing such disorders including regimens and drugs (for reducing weight) are also observed in such references.
* Unani physicians have bracketed obesity under cold derangement of temperament.
* Unani physicians have emphasized the effect of Safoof-e-Muhazzil as the main weight loss drug.
* Furthermore, Many of the drugs present in Safoof-e-Muhazzil including Lac which itself is a constituent of Safoof-e-Muhazzil have been attributed by Unani physicians to have de obstruent, desiccant, and softening and relaxant effect on vessel walls properties which further supports our hypothesis. These properties are also in cohesion with our hypothesis and perhaps these drugs may have scraping effect on atherosclerotic vessel walls.
* Lipids are metabolized mainly in the liver and it is the error of the liver or the weakness of the liver that these lipids go unchecked into the blood stream.
* Since most of constituents of Safoof-e-Muhazzil including Lac have been attributed to be liver strengthening agents, hence, due to their corrective effect on liver may help correcting raised lipid levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 Year(s) To 70 Year(s)
* Gender Both
* participate in Clinical Trial voluntarily.
* Hyperlipidemic

Exclusion Criteria:

* Persons below 20 yrs and Above 70 yrs of age
* Pregnancy
* Liver diseases
* Renal diseases
* Diabetes mellitus Type II
* Alcoholic
* AIDS
* Thyroid Disease
* Drug intake ? Corticosteroids, Diuretics, Beta-blockers, Oral contraceptives, Cyclosporin, Androgens & Retinoids

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol (TC) | six weeks
Low density Lipoprotein (LDL) | six weeks
Triglycerides (TG) | six weeks
High Density Lipoprotein (HDL) | six weeks
Very Low Density Lipoprotein (VLDL) | six weeks

SECONDARY OUTCOMES:
Waist to Hip ratio | six weeks
Body Mass Index | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Umar Jahangir, MD Scholar, Principal Investigator — Jamia Hamdard; Asim Ali Khan, MD, Principal Investigator — Jamia Hamdard
Locations (1):
- Majeedia Hospital, New Delhi, National Capital Territory of Delhi, India